CLINICAL TRIAL: NCT04768348
Title: A Prospective Study Investigating the Natural History of Adults With Phenylketonuria (PKU) Due to Phenylalanine Hydroxylase Deficiency
Brief Title: Natural History Clinical Study in Adult PKU
Status: Terminated | Type: Observational
Why Stopped: Homology Medicines has discontinued the development of this program.
Sponsor: Homology Medicines, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: HMI-100-002
Record Dates: First submitted 2021-02-18; First posted 2021-02-24 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Phenylketonurias; PKU
MeSH Terms: conditions — Phenylketonurias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of this study is to characterize the natural history of phenylketonuria (PKU) due to phenylalanine hydroxylase (PAH) deficiency in adults through prospective collection of clinical, cognitive, and quality of life assessments.

DETAILED DESCRIPTION:
Phenylalanine hydroxylase (PAH) deficiency is a rare disease caused by an inborn error of metabolism. If left untreated, PAH deficiency results in progressive, irreversible neurological impairment during infancy and early childhood.

This study is designed to collect information about important PKU-related symptoms and tests to characterize the natural history of PKU due to PAH deficiency in a selected sample of adults. No new investigational treatment will be administered to participating patients.

ELIGIBILITY:
Key Inclusion Criteria:

* Aged 18-55 years at the time of informed consent
* Diagnosis of PKU due to PAH deficiency
* One plasma Phe value with a concentration of ≥ 600 μmol/L drawn at Screening and at least 1 historical Phe value ≥ 600 μmol/L in the preceding 12 months

Key Exclusion Criteria:

* Subjects with PKU that is not due to PAH deficiency
* Alanine aminotransferase (ALT) > 1.5x upper limit of normal (ULN) and aspartate aminotransferase (AST) >1.5x ULN
* Alkaline phosphatase > 1.5x ULN
* Total bilirubin > 1.5x ULN, direct bilirubin ≥ 1.5x ULN, unless associated with Gilbert's syndrome.
* Serum creatinine > 1.5x ULN
* Hematology values outside of the normal range (hemoglobin < 11.0 g/dL for males or < 10.0 g/dL for females; white blood cells (WBC) < 3,000/μL; absolute neutrophils < 1,500/μL; platelets < 100,000/μL)
* Hemoglobin A1c > 6.5% or fasting glucose > 126 mg/dL
* Any clinically significant abnormal laboratory result at Screening, as determined by the Investigator

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Adults with diagnosed PKU due to PAH deficiency
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2021-04-20 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Plasma phenylalanine (Phe) concentrations | Baseline to Week 52
  Change in plasma Phe concentrations throughout study duration
Plasma tyrosine (Tyr) concentrations | Baseline to Week 52
  Change in plasma Tyr concentrations throughout study duration
Quality of life (QOL), as assessed using the PKU-QOL questionnaire measures | Baseline to Week 52
  Changes in PKU-QOL

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - University of South Florida, Tampa, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Community Health Clinic, Topeka, Indiana
  - University of Pittsburgh Medical Center- CHOP, Pittsburgh, Pennsylvania
  - UT Southwestern Medical Center, Dallas, Texas
  - University of Utah Health, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No